CLINICAL TRIAL: NCT04222634
Title: Metastasis-directed Therapy in Castration-refractory Prostate Cancer MEDCARE : a Non-randomized Phase 2 Trial
Brief Title: Metastasis-directed Therapy in Castration-refractory Prostate Cancer
Acronym: MEDCARE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S63177
Record Dates: First submitted 2019-12-18; First posted 2020-01-10 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Castration-resistant Prostate Cancer
MeSH Terms: interventions — Radiotherapy; Radiosurgery; Metastasectomy

STUDY DESIGN:
Intervention Model Description: single arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MDT for oligoprogressive lesions in CRPC (Other): metastasis-directed therapy:
  * radiotherapy (SBRT or conventional radiotherapy in case of local recurrence or untreated primary tumor)
  * metastasectomy
  * salvage lymphadenectomy
  * salvage prostatectomy in case of local recurrence or untreated primary tumor
  Interventions: Other: Radiotherapy (SBRT) and/or surgery (metastasectomy)

INTERVENTIONS:
Other: Radiotherapy (SBRT) and/or surgery (metastasectomy) — Metastasis-directed therapy (surgery and/or radiotherapy) as treatment for oligoprogressive lesions

SUMMARY:
The aim is to define the postponement of next line systemic treatment (NEST), by the use of metastasis-directed therapy in patients with oligoprogressive castration-refractory prostate cancer. This will be defined by the NEST-free survival.

Furthermore the investigators will use 18F PSMA PET-CT as investigational imaging, to assess the predictive value and impact on treatment policy.

DETAILED DESCRIPTION:
When treatment with pADT is initiated in case of mHSPC, the sensitivity to castration will eventually disappear due to the out-selection of castration-refractory clones. At that moment, the stage of mCRPC is attained. In the setting of mCRPC, clinical and iconographic progression (and to a lesser extent biochemical progression) traditionally implies a switch to a next-line systemic treatment (NEST). However, within the group of these progressive patients, there is a subgroup showing oligoprogressive disease, which is defined as the progression of a limited number of metastatic spots, whereas the majority of metastases is controlled by the systemic therapy the patient is receiving at that time. This heterogeneous response to treatment reflects the heterogeneity of the clonogenic cells that give rise to mCRPC. The hypothesis of this trial is that treatment with MDT of these oligoprogressive lesions allow patients to remain on their current systemic therapy, thereby delaying the need for NEST.

A multicentric retrospective chart analysis on MDT for oligoprogressive CRPC has been conductedat previously the UZ Leuven together with UZ Gent (doi: 10.1016/j.euo.2019.08.012.). A total of 30 patients with oligoprogressive CRPC were selected for further analysis. In this population, after a median follow-up of 17 months (IQR 9;25), the median NEST-FS in the MDT group was 16 months (95% CI: 10-22 months). The median progression free survival (PFS) was 10 months (95% CI: 6-15 months). Subsequently, the investigators selected within the MDT group those cases who received SBRT or surgery (metastasectomy), as these patients will be the subjects in this phase 2 trial. There was a median NEST-free survival of 21 months (CI 95% 12-21 months) and a median PFS of 10 months (95% CI: 6-14 months). SBRT or surgery-related toxicity was minor, with limited grade 1 and 2 toxicity and only one patient experiencing late grade 3 GU/GI toxicity after treatment for local relapse in the prostate.

These findings of this retrospective analysis clearly show the need for further prospective investigation. Therefore, this prospective phase 2 trial was initiated in patients with oligoprogressive mCRPC who will receive MDT. If the primary tumor has not been treated yet, local treatment will be added. Ongoing systemic treatment will be continued until progression. The trial is explorative and still hypothesis generating. The results from this trial will serve as a guidance for a randomized phase 3 trial in the near future.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven initial diagnosis of adenocarcinoma of the prostate
* mCRPC setting, with testosterone level < 50 ng/dl or 1.7 nmol/l
* Oligoprogressive disease, defined as a maximum of 3 extracranial metastases in any organ system OR local recurrence, diagnosed on conventional imaging with CT and bone scan. This may present as either the progression of pre-existing disease, and/or the appearance of new metastases. (defined according to the PCWG 3 criteria (20), see section 6. Trial Procedures)
* Patients currently treated with ADT, whether or not combined with another systemic treatment such as abiraterone acetate, enzalutamide, docetaxel and radium-223. Denosumab is allowed but not considered as second-line systemic treatment.
* Priory treated primary tumor by radiotherapy or surgery. If the primary tumour is not treated, local therapy should be added to the treatment. Both radiotherapy as well as surgery are allowed.
* WHO performance status 0-1
* Age >= 18 years old
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and/or follow-up schedule. Those conditions should be discussed with the patient before registration in the trial.
* Patient presented at the multidisciplinary tumour board of the local hospital.
* Before patient registration/randomization, written informed consent must be given according to ICH/GCO and national/local regulations.

Exclusion Criteria:

* Serum testosterone level > 50 ng/ml or > 1.7 nmol/l.
* Presence of polyprogression, defined as more than 3 progressive/new metastatic lesions and/or local recurrence (which counts for 1 lesion).
* Active malignancy other than prostate cancer that can potentially interfere with the interpretation of the trial.
* Previous treatments (RT, surgery) or comorbidities rendering PDT impossible.
* Disorder precluding understanding of trial information or informed consent or signing informed consent.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male -> prostate
Enrollment: 18 (Estimated)
Dates: Start 2019-12-27 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2030-01-01 (Estimated)

PRIMARY OUTCOMES:
Next-line Systemic Treatment - free survival (NEST-FS) | up to 5 years after MDT
  Time until the start with a subsequent systemic treatment line calculated from the last day of MDT until the first day of NEST or death (whichever comes first)
PSMA PET-CT accuracy and predictive value | up to 5 years after MDT
  We will evaluate if (1) at time of PSA progression, new lesions will be visible on PSMA PET-CT and not on conventional imaging or visible on both, (2) if those new lesions at time of radiographic progression were already visible as active lesions on PSMA PET-CT (and not on conventional imaging) at time of inclusion, and (3) we will evaluate if active lesions visible at PSMA PET-CT at initial diagnosis of oligoprogression/at time of inclusion, who are not visible on conventional imaging might disappear without targetet treatment. We will evaluate if PSMA PET-CT would result in a change of patient management.

SECONDARY OUTCOMES:
PSA response | up to 5 years after MDT
  A decline in PSA value ≥ 50% from baseline confirmed by a second value ≥ 4 weeks. Individual PSA change responses as a percentage change from baseline to week 12 will be plotted in a waterfall plot.
Clinical progression-free survival (cPFS) | up to 5 years after MDT
  Progression is defined as the appearance of any recurrence (local, nodal or metastatic) on conventional imaging.
Cancer-specific survival (CSS) | up to 10 years after MDT
  CSS is calculated from last day of treatment until PCa death
Overall survival (OS) | up to 10 years after MDT
  Overall survival (OS) will be calculated from last day of treatment until death from any cause.
Acute and late toxicity (in case of radiotherapy) | up to 5 years after MDT
  Acute and late toxicity as a result of radiotherapy will be scored using the Common Toxicity Criteria Version 5.0 (24).
Surgical complications (in case of surgery) | up to 5 years after MDT
  Surgical complications will be scored using Clavien-Dindo Classification (25) Toxicity will be scored at every follow-up visit.
Quality-of-life (QOL) | up to 5 years after MDT
  Quality of life scoring using the EORTC QLQ-30 supplemented with QLQ-PR25. We will assess the quality-of-life-years with the EuroQOL classification system (EQ-5D). Assessments are planned at baseline, last day of treatment, and during every follow-up consultation.

CONTACTS AND LOCATIONS:
Overall Officials: Gert De Meerleer, Ph.D., M.D., Principal Investigator — UZ Leuven
Locations (1):
- Gert De Meerleer, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No
Participant data will be coded and available for the involved researcher and PI only (dr. Charlien Berghen and prof. dr. De Meerleer Gert)

REFERENCES:
- [Derived] Berghen C, Joniau S, Rans K, Devos G, Poels K, Slabbaert K, Dumez H, Albersen M, Goffin K, Haustermans K, De Meerleer G. Metastasis-directed therapy in castration-refractory prostate cancer (MEDCARE): a non-randomized phase 2 trial. BMC Cancer. 2020 May 24;20(1):457. doi: 10.1186/s12885-020-06853-x. PMID 32448171